CLINICAL TRIAL: NCT06126705
Title: 18F-AlF-FAPi-04 PET/CT Imaging in Patients With Solid Tumor
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TRX0109001
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients who are surgically resectable or borderline surgically resectable plan to undergo primary lesion resection and peripheral lymph node dissection, and suspect the presence of peripheral lymph nodes or distant metastasis; Pathological results of postoperative primary lesion and lymph node dissection can be obtained
  Interventions: Drug: Radiation: 18F-AlF-FAPi-04; Drug: Radiation: 18F-FDG
- Group B (Experimental): For patients diagnosed or suspected of postoperative recurrence or late metastasis through routine imaging examination, there is at least one measurable lesion (with a short diameter of ≥ 1.5cm for lymph node lesions and ≥ 1cm for non lymph node lesions); Patients who can undergo imaging follow-up for 3-6 months or undergo pathological biopsy and puncture.
  Interventions: Drug: Radiation: 18F-AlF-FAPi-04; Drug: Radiation: 18F-FDG

INTERVENTIONS:
Drug: Radiation: 18F-AlF-FAPi-04 — Subjects who meet all the inclusion criteria will receive intravenous administration of 18F-AlF-FAPi-04 with a dosage range of 0.1-0.2 mCi/Kg. After administration, PET/CT scans will be performed at three time points: 1h, 2h, and 4h post dose. The subjects will also receive administration of 18F-FDG and undergo PET/CT scans for self-control analysis.
Drug: Radiation: 18F-FDG — Subjects who meet all the inclusion criteria will receive intravenous administration of 18F-AlF-FAPi-04 with a dosage range of 0.1-0.2 mCi/Kg. After administration, PET/CT scans will be performed at three time points: 1h, 2h, and 4h post dose. The subjects will also receive administration of 18F-FDG and undergo PET/CT scans for self-control analysis.

SUMMARY:
To evaluate the potential usefulness of 18F-AlF-FAPi-04 PET/CT for the diagnosis of primary and metastatic lesions in solid cancer.

DETAILED DESCRIPTION:
This is a prospective, single-center, two arms, open label, non-randomized study to evaluate the ability of 18F-AlF-FAPi-04 to detect FAP expressing cells in patients with solid tumor, evaluate its biological distribution characteristics, impact on clinical treatment plans, and evaluate imaging differences between different probes. Taking histopathology and imaging follow-up as gold standard, the sensitivity, specificity, and accuracy of 18F-AlF-FAPi-04 PET/CT will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain/sign informed consent.
2. Age ≥18 years, male or female patients.
3. Histologically or cytologically confirmed digestive tumors, head and neck squamous cell carcinoma, or peritoneal metastases.
4. Cohort 1: Patients with operable or borderline operable resection, scheduled for primary lesion resection and peripheral lymph node dissection, and suspected presence of peripheral lymph node or distant metastasis; The pathological results of the primary lesion and lymph node dissection were obtained.

   Cohort 2: Patients with confirmed or suspected postoperative recurrence or advanced metastasis by routine imaging had at least one measurable lesion; Patients who can undergo imaging follow-up for 3 to 6 months or can undergo pathological biopsy.
5. The ECOG score is 0-2
6. Patients with adequate organ function.

Exclusion Criteria:

1. Previously received FAP-targeted radioligand therapy.
2. Patients are participating in any other clinical trials or receiving investigational drugs.
3. Patients with central nervous system (CNS) metastases with symptoms or receiving glucocorticoid therapy to maintain functional integrity of the nervous system.
4. Patients with other malignancies that may interfere with disease assessment, who have a prior history of malignancy but have been adequately treated, who have not been treated for more than 3 years prior to enrollment, and who have no evidence of recurrence are eligible to participate in the study.
5. Comorbidities with serious or poorly controlled medical conditions, including but not limited to hard-to-control infections, known active hepatitis B or C, or other conditions that investigators believe may impair study participation or collaboration.
6. A physical or psychiatric history that may interfere with the purpose and evaluation of the study, or any condition in which the investigator determines that the patient is incapable of cooperating with imaging and procedures.
7. Patients who do not consent to effective contraception or restricted sexual practices.
8. There are other conditions that the investigator deems unsuitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Group A: Sensitivity and Specificity of 18F-AlF-FAPi-04 | 6 months after last dose administration
  Performance [sensitivity, specificity, accuracy] of 18F-AlF-FAPi-04 PET imaging to detect FAP-expressing cells, using surgical histopathological results as truth standard
Group B: Sensitivity and Specificity of 18F-AlF-FAPi-04 | 6 months after last dose administration
  Performance [sensitivity, specificity, accuracy] of 18F-AlF-FAPi-04 PET imaging to detect FAP-expressing cells, using imaging follow-up or histopathological puncture results as truth standard

SECONDARY OUTCOMES:
Biodistribution of 18F-AlF-FAPi-04 | 120 minutes after tracer injection
  The biodistribution of 18F-AlF-FAPi-04 in normal and cancer tissues of patients with various malignancies will be measured by average and maximum standardized uptake value (SUVmean and SUVmax)

CONTACTS AND LOCATIONS:
Overall Officials: Huang xiaohong, MM, Principal Investigator — Afﬁliated Hospital of North Sichuan Medical College
Locations (1):
- Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: No